CLINICAL TRIAL: NCT05980455
Title: Randomized Study of Enterra Programming with Nocturnal Cycling in Gastroparetics
Brief Title: Study of Enterra Programming with Nocturnal Cycling in Gastroparetics
Acronym: RESTING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Enterra Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLN 001-PR-00755
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Gastroparesis; Gastroparesis Nondiabetic; Gastroparesis Due to Diabetes Mellitus
Keywords: Gastric electrical stimulation; Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Control Sleep Cycle (Active Comparator): Baseline device programming parameters will be used during study participation. No modification to Enterra® device programming will be in effect during waking or sleeping hours.
  Interventions: Device: Enterra® Therapy System
- Arm 1 Sleep Cycle (Experimental): Device programming parameters participants have at enrollment will be used during waking hours.
  During sleeping hours, the Enterra® device will cycle through modified programming over the course of 6 hours. Each hour, the Enterra® device will deliver 30 minutes of reduced stimulation, followed by 30 minutes of waking hours stimulation. At the end of the 6-hour sleep cycle, the Enterra® device will return to waking hours programming.
  Interventions: Device: Enterra® Therapy System
- Arm 2 Sleep Cycle (Experimental): Device programming parameters participants have at enrollment will be used during waking hours.
  During sleeping hours, the Enterra® device will cycle through modified programming over the course of 8 hours. Each hour, the Enterra® device will deliver 45 minutes of reduced stimulation, followed by 15 minutes of waking hours stimulation. At the end of the 8-hour sleep cycle, the Enterra® device will return to waking hours programming.
  Interventions: Device: Enterra® Therapy System

INTERVENTIONS:
Device: Enterra® Therapy System — The Enterra® Therapy System for gastric electrical stimulation (GES) is indicated for the treatment of chronic intractable (drug refractory) nausea and vomiting secondary to gastroparesis of diabetic or idiopathic etiology in patients aged 18 to 70 years.
  Other Names: Gastric electrical stimulation

SUMMARY:
The purpose of this research study is to evaluate if different Enterra® device programming methods active during sleeping hours can maintain gastroparesis-related symptom relief and quality of life measures.

Participants in this study with existing Enterra® devices will be randomly assigned to one of three programming methods that will be active during sleep. Participants will answer daily questions about their gastroparesis symptoms on an application with their phone/tablet. Participants will answer quality of life questionnaires about their gastroparesis symptoms at study visits.

Participants will be involved in the study for up to six months after treatment assignment.

Programming parameters in the study are within currently approved labeling.

ELIGIBILITY:
In order to be eligible to participate in this study, a participant must meet all of the following criteria:

1. Completed informed consent process with signed and dated informed consent form;
2. Stated willingness to comply with all study procedures and availability for the duration of the study;
3. Male or female, aged ≥18 or ≤70 at time of informed consent;
4. Currently implanted with the Enterra® Therapy System (Enterra® II 37800 neurostimulator);
5. High GES output defined as remaining pulse generator expected life of > 9 months from enrollment and less than 4 years from the time of implant;
6. Stable gastroparesis symptoms, in the opinion of the investigator;
7. On stable medical therapy for gastroparesis symptoms;
8. On stable supplemental nutritional support during the month prior to enrollment;
9. English language comprehension to complete study-required assessments;
10. Reliable access to internet-connected smart device(s) to complete study-required assessments.

A participant who meets any of the following criteria will be excluded from participation in this study:

1. Post-surgical gastroparesis (e.g., fundoplication, Bilroth I or II) or other active stomach or gastrointestinal diseases disorders which could explain symptoms in the opinion of the investigator;
2. Subjects, in the opinion of the investigator, with profound nausea and/or vomiting at night;
3. Subjects, in the opinion of the investigator, with profound gastroparesis symptoms upon waking in the morning;
4. Subjects without a regular and defined sleep schedule;
5. Pregnancy, or subject that intends to become pregnant during participation in the study;
6. Chemical dependency;
7. Enterra lead impedance measurements ≥ 700 Ohms at screening visit;
8. Life expectancy < 1 year from conditions other than GI diseases;
9. Subjects with an underlying disease leading to follow-up by MRI outside of current MR conditional indications;
10. Participation in other clinical studies;
11. Subjects involved in current or past medical-related litigation;
12. Subjects with cognitive impairment or other characteristic that would limit subject's ability to complete study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Weekly Vomiting Frequency by GCSI-DD | 3 Months, 6 Months
  Less than a 50% increase in GCSI-DD weekly vomiting frequency from baseline
Scoring Change in Nausea Severity by GCSI-DD | 3 Months, 6 Months
  Less than a 1-point increase in GCSI-DD nausea severity from baseline

SECONDARY OUTCOMES:
Mean Change from Baseline in GCSI-DD Total Symptom Score | 3 Months, 6 Months
  Change in GCSI-DD Total Symptom Score from baseline
Mean Change from Baseline in GCSI-DD Nausea Severity | 3 Months, 6 Months
  Change in GCSI-DD nausea severity from baseline
Mean Change from Baseline in GCSI-DD Weekly Vomiting Frequency | 3 Months, 6 Months
  Change in GCSI-DD weekly vomiting frequency from baseline
Mean Change from Baseline in PAGI-QoL Scores | 3 Months, 6 Months
  Change in PAGI-QoL from baseline
Mean Change from Baseline in Quality of Sleep Scores | 3 Months, 6 Months
  Change in Quality of Sleep from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Stocker, MD, Principal Investigator — University of Louisville
Locations (2):
- United States (2):
  - University of Louisville, Louisville, Kentucky
  - MNGI Digestive Health, P.A., Coon Rapids, Minnesota

IPD SHARING:
Plan to Share IPD: No